CLINICAL TRIAL: NCT01166763
Title: Modulation of Breast Cancer Risk Biomarkers by High Dose Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: BTR Group (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11657
Record Dates: First submitted 2010-07-16; First posted 2010-07-21 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: breast atypia; high risk for breast cancer; random periareolar fine needle aspiration; RPFNA; breast epithelial hyperplasia; ki-67; chemoprevention; vitamin D3; Additional relevant MeSH terms:; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs; Breast Neoplasms; Pharmacologic Actions; Hyperplasia; high risk for development of breast cancer; Neoplasms; Neoplasms by Site; Pathologic Processes; Antirheumatic Agents; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Hyperplasia; Neoplasms; Neoplasms by Site; Pathologic Processes; Breast Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high dose vitamin D3 (10,000 IU weekly) (Experimental): Group/Cohort Label vitamin D3
  Interventions: Drug: vitamin D3

INTERVENTIONS:
Drug: vitamin D3 — oral capsules, 10,000 IU per week for 6 months
  Other Names: Maximum D3

SUMMARY:
The overall goal of this project is to determine if high dose vitamin D3 given to premenopausal women at high risk for development of breast cancer, who initially have insufficient levels of 25-hydroxy vitamin D (<30 ng/ml), will raise 25(OH)D levels above 50 ng/ml. If so, will certain risk biomarkers for development of breast cancer be reliably and favorably modulated?

DETAILED DESCRIPTION:
Protocol Objectives:

To determine if high dose vitamin D3 given to premenopausal women who initially have insufficient levels of 25-hydroxy vitamin D (<30 ng/ml) will raise 25(OH)D levels above the 50 ng/ml level considered to be required for breast health. If so, will certain risk biomarkers for development of breast cancer be reliably and favorably modulated? The primary endpoint will be a decrease in mammographic breast density (percent area considered at increased density). Change in proliferation (a decrease as assessed by Ki-67) will also be examined. Modulate of expression of genes important in breast cancer risk or reflective of vitamin D's mechanism of action will be studied using quantitative real time polymerase chain reaction (qRT-PCR).

Study Design:

The study is a single-arm open label clinical trial. Women who are high risk for development of breast cancer on the basis of family or personal history will undergo random periareolar fine needle aspiration (RPFNA) to acquire breast cells for assessment of gene expression by qRT-PCR. Women with mammographic density >10% will be eligible for enrollment. All subjects will receive high dose vitamin D3 (3 capsules of 10,000 IU of vitamin D3 every week for 6-8 months). At that time, a repeat RPFNA and mammogram will be performed. Measurement of serum levels of 25(OH)D will be performed at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be premenopausal women age 55 or younger, and actively menstruating with 4 or more periods per year.
* Subjects may be using barrier contraceptive, an intrauterine device, a Nuvaring, or similar non-oral contraceptive; or oral contraceptives.
* Subjects must be at increased risk for breast cancer on the basis of at least one of the following criteria:

  * five-year Gail risk of 3X the average risk of the age group;
  * a first degree relative with breast cancer under the age of 60 or multiple second degree relatives with breast cancer;
  * prior biopsy exhibiting atypical hyperplasia (AH), LCIS, DCIS, RPFNA evidence of hyperplasia with atypia within the last three years;
  * Chest or neck radiation before age 30;
  * Breast density equals or exceeds 50 percent.
* If previously on a chemoprevention agent or prevention trial, subjects must have completed study participation at least 6 months prior to baseline biomarker assessment.
* If subject has a history of AH, LCIS, or ER-positive DCIS by diagnostic biopsy, must have been counseled about appropriate standard prevention therapies such as tamoxifen and is either not eligible or is not interested in standard prevention therapies. Women with DCIS must have had appropriate local therapy (lumpectomy plus radiation or mastectomy).
* Subject must have had a mammogram performed at the University of Kansas Breast Imaging Center with estimated visual breast density of greater than 10 percent.
* Subject must have had within six months prior to entering the study, an RPFNA during the follicular portion (day 1-10) of the menstrual cycle with material for cytomorphology, Ki-67 and qRT-PCR; in addition to serum obtained and banked.
* Subjects must have 25(OH)D level < 30 ng/ml as measured within 8 weeks of starting intervention. Subjects may have been identified as having low vitamin D levels through participation in HSC 11313, Osteopenia/Osteoporosis in Pre-menopausal Women at High Risk for Development of Breast Cancer, but low level must be confirmed within 8 weeks prior to starting study agent Subject must be willing to continue the same hormonal milieu present at baseline throughout trial.
* Subjects must be willing to undergo measurement of height, weight, and BMI at initiation of intervention.
* Subjects must have participated in HSC 11313, and have had a DEXA scan for bone density and body fat analysis on the GE Lunar Prodigy Advance research unit in the Breast Cancer Survivorship Center.
* Subjects must be willing to sign an informed consent for the entire study and separate consent for repeat RPFNA.

Exclusion Criteria:

* Women that have had a metastatic malignancy of any kind.
* Women that have had prior invasive breast cancer If subject has had a DCIS, at least two months must have elapsed from surgery and/or radiation therapy to the involved breast. Only the contra-lateral (uninvolved breast) will be studied by FNA. The subject may not have had any radiation therapy to the contra-lateral breast to be studied.
* Women who are pregnant or nursing.
* Women who have taken a SERM, aromatase inhibitor or participated in a chemoprevention or other investigational drug study within six months prior to baseline FNA.
* Women who have used fertility drugs within six months prior to baseline aspiration.
* Women with a history of sarcoidosis, hypercalcemia, hyperparathyroidism, or renal stones.
* Women who are receiving treatment for rheumatoid arthritis or other connective tissue diseases.
* Women who have an elevated blood calcium level at baseline; defined as any elevation above the institutional normal range.

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Global results only will be published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment April 2009 to December 2010. Breast Cancer Prevetnion Center at University of Kansas Medical Center
Period: Overall Study
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Started | 30
Completed | 27
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (4.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Gail Risk 5-year Probability of Cancer Development [Mean (Standard Deviation); unit: percent probability] — Gail model is an algorithm to calculate a predicted probability of developing breast cancer within the next 5 years.
  percent probability | 1.6 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mammographic Breast Density Over Course of Study
Description: Change in the percent of the breast area that is considered to be at higher density on mammogram.
Time Frame: baseline and 6 months
Population: All subjects completing trial
Measure: Mean (Standard Deviation); unit: Change in percent dense breast area
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Number analyzed (Participants) | 27
Change in percent dense breast area | -0.5 (5.8)

2. Secondary Outcome: Change in Proliferation (as Assessed by Ki-67) Examined in Breast Epithelial Cells.
Description: Change in percent of cells expressing staining for Ki-67 antibody in breast epithelial cell specimens acquird by Random Periareolar Fine Needle Aspiration.
Time Frame: baseline and 6 months
Population: All subjects completing trial.
Measure: Median (Full Range); unit: percentage of cells staining positive
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Number analyzed (Participants) | 27
percentage of cells staining positive | -0.4 [-4.0 to 4.8]

3. Secondary Outcome: OH Vitamin D Levels in Serum
Description: Assessment of 25(OH)D levels as a measure of circulating vitamin D.
Time Frame: baseline and 6 months
Population: All subjects completing trial
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Number analyzed (Participants) | 27
ng/ml | 55.4 (13.8)

ADVERSE EVENTS:
Time Frame: 6 months duration of study agent administration
Arm/Group | High Dose Vitamin D3 (10,000 IU Weekly)
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D3 (10,000 IU Weekly) (N=30)
Cholecystitis (Gastrointestinal disorders) | 1 (1) — Grade 3, considered not to be related to study agent.
Flank pain (Nervous system disorders) | 1 (1) — Grade 3 flank pain, not considered to be related to study agent
Increase in diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3, not considered to be related to study agent.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D3 (10,000 IU Weekly) (N=30)
Headache (Nervous system disorders) | 2 (30) — Grade 2 headache
Abdominal cramps (Gastrointestinal disorders) | 1 (2) — Grade 2 (2 instances in same subject)

LIMITATIONS AND CAVEATS:
Single arm pilot trial so all comparisons are within subject for change over the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes